CLINICAL TRIAL: NCT06785428
Title: Dietary Protein Requirements in Adults With Facioscapulohumeral Muscular Dystrophy
Acronym: FSHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A06-M33-23B
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Fascioscapulohumeral Muscular Dystrophy
Keywords: Protein requirements; Facioscapulohumeral muscular dystrophy; Indicator amino acid oxidation technique
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with FSHD (Experimental): Participants are to be randomly assigned varying levels of amino acid intakes ranging between 0.2 to 2.8 g/kg/d.
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Amino acid intakes will vary between 0.2 to 2.8 g/kg/d.

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is one of the most common types of muscular dystrophy, affecting about 4 out of 100,000 individuals. The disease is characterized by progressive muscle loss (i.e., muscle atrophy) commonly affecting the face, shoulders, and upper arm muscles. The muscle loss ultimately results in reduced strength and impaired physical performance. At present there is no cure for FSHD, therefore, physicians have focused on therapeutic interventions to help alleviate these symptoms.

Daily consumption of adequate amounts of dietary protein is essential to support muscle mass maintenance and overall health and function across the lifespan. However, previous research has reported inadequate protein intake in individuals with FSHD. The characteristic of progressive muscle loss in individuals with FSHD and other muscular dystrophies is ultimately due to an imbalance in the rate of muscle building (i.e., muscle protein synthesis) and muscle breakdown (i.e., muscle protein breakdown), where individuals with FSHD have been shown to have reduced rates of muscle building. As inadequate protein intake is known to result in a loss of muscle mass, strength and function, this loss may be amplified in individuals with FSHD.

Dietary recommendations traditionally have been determined through nitrogen balance techniques, where the current recommended dietary allowance (RDA) for daily protein intake for adults is 0.8 g/kg/d. However, recent research indicates how the nitrogen balance technique potentially underestimates protein requirements. Therefore, there is a need to reassess current dietary recommendations in adults with FSHD in order to help support the maintenance of muscle strength and function.

Recent efforts to understand protein requirements in various populations have been completed using the indicator amino acid oxidation technique (IAAO). This non-invasive method is reported to provide a robust measure of protein requirements. Due to its non-invasive nature, the IAAO method allows researchers to use this technique in individuals with FSHD, where there is currently limited work in studying this population.

The purpose of this study is to measure the protein requirements in individuals with FSHD using the non-invasive IAAO technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male participants who are 26 to 60 years of age at screening (inclusive)
* Genetically confirmed with FSHD
* Ambulatory
* Has maintained stable use of medication and supplements, stable dietary and lifestyle habits, and stable body weight, for the last 3 months prior to screening and agree to maintain them throughout the study
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures

Exclusion Criteria:

* Individuals who are lactating or pregnant
* Usage of corticosteroids within 3 months of study entry or had ever taken steroids for a duration exceeding 1 year
* On androgens or growth hormone within 6 months before screening and for duration of study; topical physiologic androgen replacement is permitted
* On sympathomimetic agents, antidepressants, or β-receptor blockers
* Have cardiovascular disease
* Evidence of an alternative diagnosis other than FSHD or a coexisting myopathy or dystrophy
* Current/active malignancy (e.g., remission less than 5 years' duration), with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
* Type 1 or type 2 diabetes mellitus
* History of sensitivity to protein pharmaceuticals
* Known active substance abuse, including alcohol
* Renal impairment (serum creatinine ≥ 2 times the upper limit of normal,(ULN))
* History of severe restrictive or obstructive lung disease, or evidence for interstitial lung disease on screening chest radiograph
* Major surgery within 4 weeks prior to metabolic trial 1
* Any other active or unstable medical/psychological conditions or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
13CO2 Excretion | 7-weeks
  Measured by continuous-flow isotope ratio mass spectrometry

SECONDARY OUTCOMES:
L-[13C]-Phenylalanine Oxidation | 7-weeks
  Measured by gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- McGill university, Montreal, Quebec, Canada